CLINICAL TRIAL: NCT05902143
Title: Evaluation of Fine Motor Function in Children With Specific Learning Disorders
Brief Title: Fine Motor Function in Children With Specific Learning Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, Assoc. Prof. PhD, Akdeniz University
Other Study IDs: 2022-297
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Specific Learning Disorder
Keywords: Specific Learning Disorder; Fine motor skills; Grip strength; Upper extremity; Children
MeSH Terms: conditions — Specific Learning Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: children with Specific Learning Disorder
- Control Group: children with typically developing children

SUMMARY:
Specific Learning Disorder (SLD) is a neurodevelopmental disorder in which a person shows difficulties in reading, written narration, and/or mathematics. 30 to 50 percent of children with SLD experience difficulties in fine motor skills, such as handwriting skills, and also during self-care activities and activities that require sorting. This study will evaluate children with SLD and healthy ages within fine motor skills, handgrip strength, and hand-forearm anthropometric measurements. Our study will show the impact of the fine motor skills of children with SLD on their quality of life and participation in daily life activities. In light of our current knowledge, no study has been found that comprehensively examines the fine motor functions of children with SLD. Therefore, normative data on the upper extremity functions of children with SLD will be presented to the literature. In this context, our work will shed light on the development of new treatments and assessment methods for clinicians and researchers working with children with SLD.

DETAILED DESCRIPTION:
Specific Learning Disorder (SLD) is a neurodevelopmental disorder in which the individual has difficulties in reading, written expression, and/or mathematics, according to the Diagnostic and Statistical Manual of Mental Disorders - 5 (DSM-V). SLD; According to DSM-5, the academic difficulties experienced are explained in detail by dividing them into three subgroups. These are dyslexia, dyscalculia, and dysgraphia. The incidence of SLD is approximately 33% in girls and 67% in boys between the ages of 6-12. The ethology of SLD is multifactorial. It is associated with multiple genes and environmental risk factors. Structural imaging studies in children with SLD have revealed that grey matter is reduced. As a result of low grey matter, early literacy education seems to be negatively affected, and fine motor skills such as writing play an important role in this influence.

Writing is a complex activity that includes perceptual, motor, and cognitive processes. Writing activities require a high level of fine motor coordination, postural control, adjustable grip strength, visual perception, and language skills. Considering the studies, it is stated that children who go to primary school spend 31%-60% of their academic days with tasks involving fine motor skills, and most of them do activities such as writing and painting. In addition to their academic and writing performances, children with SLD perform differently in daily life compared to their healthy peers. In general, they have difficulties during self-care activities such as tying shoes, clipping their nails, buttoning/zipping, shaving, and performing activities that require sequencing. At the same time, children with SLD have difficulties in sensory processing, balance, and postural control. Difficulties in sensory processing, balance, and postural control seen in children with SLD affect proximal stability. When proximal stability is poor, distal movements cannot be performed in good quality. Therefore, adequate postural control and proximal stability are essential prerequisites for many activities of daily living. In the literature, it has been shown that grip strength and anthropometric characteristics of the upper extremity affect distal fine motor skills. In a study by Anakwe et al., it was shown that grip strength increased as the forearm circumference measurement value increased. In a study examining the relationship between hand grip and finger strength and anthropometric measurements, it was concluded that grip strength increased as arm and forearm measurements increased. It has been proven that grip strength increases as arm and forearm measurements increase.

In the light of our current knowledge, no study has been found that comprehensively examines the fine motor functions, hand and finger strengths, and anthropometric measurements of children with SLD. The primary aim of this study is to examine the fine motor skills, hand grip strength, and hand and forearm anthropometric characteristics of children with SLD compared to those of healthy children and to investigate their relationships with each other. The second aim of our study is to examine the effect of fine motor skills on quality of life and participation in activities at home, school, and community environment of children with SLD compared to their healthy peers.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years old
* Patients diagnosed with SLD by a physician, regardless of subtype.
* Cognitive ability to follow instructions for assessment measures
* Families and children who agreed to participate in the study

Exclusion Criteria:

* Any psychiatric diagnosis such as autism spectrum disorder, psychotic symptoms, depression

  * Children with a neurological or orthopedic disorder such as head trauma, Cerebral Palsy, epileptic seizures and speech disorder
  * Families and children who do not agree to participate in the study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children with specific learning disorder and typically developing peers
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-02-12 (Estimated)

PRIMARY OUTCOMES:
Bruininks-Oseretsky Test of Motor Proficiency-2 (BOT-2) | Baseline
  Bruininks-Oseretsky Test of Motor Proficiency-2 (BOT-2) is norm referenced and designed to measure gross and fine motor skills in youth 4 to 21 years of age. Standard scores 40 are considered below average, whereas those >40 range from average to above average.
Purdue Pegboard Test | Baseline
  The Purdue Pegboard Test consists of a board with four subtests: Dominant hand, Non-Dominant hand, Bimanual and Assembly. Each subtest was administered three times in a row. The dominant hand and non-dominant hand subtests required to place as many pegs as possible in the column corresponding to the hand being tested within 30-sec. The dominant hand is tested first followed by the non-dominant hand. In the bimanual subtest, both hands simultaneously placed a pair of pegs in both columns. The scores on these three tests were the pairs of pegs for the bimanual subtest, placed within 30-sec. The assembly subtest required picking up and placing pegs, washers, collars and second washers using alternating hands. This score represents the number of pieces assembled within 60-sec.
Hand Dynamometer | Baseline
  Hand Dynamometer will be used to evaluate hand grip strength. Measurements will be performed in the position defined by the American Association of Hand Therapists. During the test, the child will be seated with a 90° flexion angle of the hip and knee. Three measurements will be made to measure the hand grip strength.
Pinch Gauge | Baseline
  "Pinch Gauge" will be used to evaluate finger strength. Measurements will be performed in the position defined by the American Association of Hand Therapists. Finger strengths will be recorded by asking the children to grasp at maximal strength in the three basic types of fine grip. These are fingertip grip, lateral grip, and three-point grip positions, respectively.

SECONDARY OUTCOMES:
Participation and Environment Measurement Child & Youth (PEM-CY) | Baseline
  Participation and Environment Measurement Child & Youth (PEM-CY) is a parent-report questionnaire to assess participation and environment factors in the home, at school and within community Settings. The participation sections included 10 activities in the home setting, five activities in the school setting and 10 in the community setting. For each activity, parents are asked to determine the participation frequency (how frequently has the child participated with eight options: daily to never), participation involvement (how involved the child is while participating the activity rated on a five-point scale: very involved to minimally involved) and whether change is desired (do the parents want to see change in the child's participation in this type of activity: no or yes, with 5 different types of change).
The Pediatric Quality of Life Inventory (PEDS-QL) | Baseline
  The Pediatric Quality of Life Inventory (PEDS-QL) is a generic health related quality of life measure consisting of 4 core scales, physical function (8 items), emotional function (5 items), social function (5 items) and school function (5 items) that is intended for use in healthy and patient populations. Respondents are asked to recall the last month and indicate how frequently - from never to almost always - they have experienced specific phenomena. Item responses (0-100) are averaged to form total and core scores; higher scores indicate higher functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silver CH, Ruff RM, Iverson GL, Barth JT, Broshek DK, Bush SS, Koffler SP, Reynolds CR; NAN Policy and Planning Committee. Learning disabilities: the need for neuropsychological evaluation. Arch Clin Neuropsychol. 2008 Mar;23(2):217-9. doi: 10.1016/j.acn.2007.09.006. Epub 2007 Oct 30. PMID 17977692
- [Background] Rutter M, Caspi A, Fergusson D, Horwood LJ, Goodman R, Maughan B, Moffitt TE, Meltzer H, Carroll J. Sex differences in developmental reading disability: new findings from 4 epidemiological studies. JAMA. 2004 Apr 28;291(16):2007-12. doi: 10.1001/jama.291.16.2007. PMID 15113820
- [Background] Darki F, Peyrard-Janvid M, Matsson H, Kere J, Klingberg T. Three dyslexia susceptibility genes, DYX1C1, DCDC2, and KIAA0319, affect temporo-parietal white matter structure. Biol Psychiatry. 2012 Oct 15;72(8):671-6. doi: 10.1016/j.biopsych.2012.05.008. Epub 2012 Jun 9. PMID 22683091
- [Background] Raschle NM, Chang M, Gaab N. Structural brain alterations associated with dyslexia predate reading onset. Neuroimage. 2011 Aug 1;57(3):742-9. doi: 10.1016/j.neuroimage.2010.09.055. Epub 2010 Sep 25. PMID 20884362
- [Background] Goldstand S, Gevir D, Yefet R, Maeir A. Here's How I Write-Hebrew: Psychometric Properties and Handwriting Self-Awareness Among Schoolchildren With and Without Dysgraphia. Am J Occup Ther. 2018 Sep/Oct;72(5):7205205060p1-7205205060p9. doi: 10.5014/ajot.2018.024869. PMID 30157018
- [Background] Di Brina C, Averna R, Rampoldi P, Rossetti S, Penge R. Reading and Writing Skills in Children With Specific Learning Disabilities With and Without Developmental Coordination Disorder. Motor Control. 2018 Oct 1;22(4):391-405. doi: 10.1123/mc.2016-0006. Epub 2018 Feb 28. PMID 29488824
- [Background] McHale K, Cermak SA. Fine motor activities in elementary school: preliminary findings and provisional implications for children with fine motor problems. Am J Occup Ther. 1992 Oct;46(10):898-903. doi: 10.5014/ajot.46.10.898. PMID 1463061
- [Background] Moe-Nilssen R, Helbostad JL, Talcott JB, Toennessen FE. Balance and gait in children with dyslexia. Exp Brain Res. 2003 May;150(2):237-44. doi: 10.1007/s00221-003-1450-4. Epub 2003 Apr 8. PMID 12682807
- [Background] Cowley JC, Gates DH. Inter-joint coordination changes during and after muscle fatigue. Hum Mov Sci. 2017 Dec;56(Pt B):109-118. doi: 10.1016/j.humov.2017.10.015. Epub 2017 Nov 6. PMID 29121490
- [Background] Anakwe RE, Huntley JS, McEachan JE. Grip strength and forearm circumference in a healthy population. J Hand Surg Eur Vol. 2007 Apr;32(2):203-9. doi: 10.1016/J.JHSB.2006.11.003. Epub 2007 Jan 2. PMID 17197064